CLINICAL TRIAL: NCT05411965
Title: A Randomized, Open-label, Single Dose, Two-way Crossover Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR3003" and Co-administration of "BR3003B" and "BR3003C" in Healthy Volunteers.
Brief Title: A Study to Evaluate the Pharmacokinetics After Administration of BR3003 and Co-administration of BR3003B and BR3003C.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-DPC-CT-101
Record Dates: First submitted 2022-05-26; First posted 2022-06-09 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dapagliflozin; Pioglitazone

STUDY DESIGN:
Intervention Model Description: two-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence Group A (Experimental): The investigational products will be administered according to the treatment groups assigned to each sequence group in Period 1 and Period 2.
  *Sequence A [Period 1] Co-administration of BR3003B(R1) and BR3003C(R2) (single dose)
  - Wash out for 7 days [Period 2] Administration of BR3003(T) (single dose)
  Interventions: Drug: BR3003(T); Drug: BR3003B(R1); Drug: BR3003C(R2)
- Sequence Group B (Experimental): The investigational products will be administered according to the treatment groups assigned to each sequence group in Period 1 and Period 2.
  *Sequence B [Period 1] Administration of BR3003(T) (single dose)
  - Wash out for 7 days [Period 2] Co-administration of BR3003B(R1) and BR3003C(R2) (single dose)
  Interventions: Drug: BR3003(T); Drug: BR3003B(R1); Drug: BR3003C(R2)

INTERVENTIONS:
Drug: BR3003(T) — Test drug (T):"BR3003" Boryung Pharmaceutical Co., Ltd.
  Other Names: Dapagliflozin 10mg / Pioglitazone 30mg
Drug: BR3003B(R1) — Reference drug 1 (R1): "BR3003B" of Celltrion Pharm, Inc.
  Other Names: Pioglitazone 30mg
Drug: BR3003C(R2) — Reference drug 2 (R2): "BR3003C" of AstraZeneca Korea
  Other Names: Dapagliflozin 10mg

SUMMARY:
To perform a comparative evaluation on the pharmacokinetics and the safety after administration of "BR3003" and co-administration of "BR3003B" and "BR3003C" in healthy adults.

DETAILED DESCRIPTION:
A randomized, open-label, single oral dose, two-way crossover study under fasting condition. Target number of subjects: 46 subjects in total.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are 19 years old or older at the screening visit.
2. Those whose weight is ≥50kg (≥45kg for female subjects) and their body mass index (BMI) shall be between 18.0 kg/m2 and 30.0 kg/m2.
3. Those without clinically significant congenital or chronic diseases at the screening visit and without any pathological symptom or opinion after an internal medicine examination.
4. Those who are judged eligible for the trial by the principal investigator (or an authorized trial doctor) according to diagnostic tests such as hematology test, blood chemistry test, serology test and urinalysis that are predefined according to the characteristics of the investigational drugs in addition to ECG results.
5. Those who agree to rule out the possibility of pregnancy through medically acceptable methods of contraception* used by the subject himself/herself or his/her spouse/partner from the first administration of the investigational drugs to 7 days after the last administration of the investigational drugs, and those who agree not to donate their sperms or eggs.
6. Those who are given detailed explanations about the trial objectives, components as well as the properties of the investigational drugs and express their voluntary consent to participate in the trial by signing a written consent.

Exclusion Criteria:

1. Those who currently have or have history of clinically significant diseases related to digestive system, cardiovascular system, endocrine system, respiratory system, hemato-oncology, infection, kidney and genitourinary system, neuropsychiatric system, musculoskeletal system, immune system, Ear-Nose-Throat system, dermal system, ophthalmologic system, etc.
2. Those who have medical history of gastrointestinal resection (however, appendectomy and hernia operation shall be excluded) or gastrointestinal system diseases that may influence the absorption of drugs.
3. Those who took drugs that substantially induce or inhibit drug-metabolizing enzymes of barbiturates, etc. in 30 days prior to the first administration or who took drugs that can impact the study in 10 days before the first administration. (However, subjects may participate in the study as judged by the principal investigator (or an authorized trial doctor) in consideration of pharmacokinetic or pharmacodynamic characteristics such as the interaction with the investigational drugs and half-life of co-administered drugs.)
4. Those who have participated in a bioequivalence study or other clinical trials and have been administered with investigational drugs in 180 days prior to the first administration. (The day of the last administration of investigational drugs shall be counted as day 1 of the end of trial.)
5. Those who have given a whole blood donation in 60 days prior to the first administration, who have given an apheresis blood donation in 14 days prior to the first administration or who have received blood transfusion in 30 days prior to the first administration.
6. Those who are applicable to the following conditions in 30 days prior to the first administration:

   * Male subjects: average alcohol intake > 21 units/week
   * Female subjects: average alcohol intake > 14 units/week

     (1 unit= 50 mL of soju, 30 mL of hard liquor or 250 mL of beer)
   * Daily average smoking of >20 cigarettes
7. Those who apply to the following criteria

   * Those who have medical history of hypersensitivity to major ingredients, other ingredients or additives of the investigational drugs.
   * Those who have diabetic ketoacidosis, diabetic coma and precoma or type 1 diabetes.
   * Those who are under dialysis.
   * Those who currently have or have medical history of heart failure.
   * Those who have active bladder cancer or have history of bladder cancer.
   * Those who have hepatopathy or severe renal impairment.
   * Those who have severe infection or severe trauma before or after surgery.
   * Those who have uninvestigated, gross hematuria.
   * Those who have genetic problems including galactose intolerance, Lapp lactase deficiency and glucose-galactose malabsorption.
   * Those whose eGFR is < 60 mL/min/1.73 m2.
8. Others who are judged ineligible to participate in the trial by the principal investigator (or an authorized trial doctor) due to reasons other than the above inclusion/exclusion criteria.
9. Female volunteers who are pregnant, suspected to be pregnant or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-07-03 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables - AUC | Pre-dose(0hour), 0.167hour(10 min), 0.333hour(20 min), 0.5hour(30 minutes), 0.667hour(40min), 1hour, 1.5hour, 2hour, 3hour, 4hour, 5hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  Area under the plasma concentration versus time curve(AUCt) of Pioglitazone and Dapagliflozin(Blood samples are collected 22 times for each Period.)
Pharmacokinetic variables - Cmax | Pre-dose(0hour), 0.167hour(10 min), 0.333hour(20 min), 0.5hour(30 minutes), 0.667hour(40min), 1hour, 1.5hour, 2hour, 3hour, 4hour, 5hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  Peak Plasma Concentration(Cmax) of Pioglitazone and Dapagliflozin(Blood samples are collected 22 times for each Period.)

SECONDARY OUTCOMES:
Pharmacokinetic variables - AUC∞ | Pre-dose (0hour), 0.167hour (10min), 0.333hour (20 min), 0.5hour (30 min), 0.667hour (40min), 1hour, 1.5hour, 2hour, 3hour, 4hour, 5hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  AUC∞ of Pioglitazone and Dapagliflozin (Blood samples are collected 22 times for each Period.)
Pharmacokinetic variables - AUCt/AUC∞ | Pre-dose (0hour), 2hour, 4hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  AUCt/AUC∞ of Pioglitazone and Dapagliflozin (Blood samples are collected 22 times for each Period.)
Pharmacokinetic variables - Tmax | Pre-dose (0hour), 0.167hour (10min), 0.333hour (20 min), 0.5hour (30 min), 0.667hour (40min), 1hour, 1.5hour, 2hour, 3hour, 4hour, 5hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  Tmax of Pioglitazone and Dapagliflozin (Blood samples are collected 22 times for eachour Period.)
Pharmacokinetic variables - t1/2 | Pre-dose (0hour), 0.167hour (10min), 0.333hour (20 min), 0.5hour (30 min), 0.667hour (40min), 1hour, 1.5hour, 2hour, 3hour, 4hour, 5hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  t1/2 of Pioglitazone and Dapagliflozin (Blood samples are collected 22 times for eachour Period.)
Pharmacokinetic variables - AUCt of Pioglitazone M-IV | Pre-dose (0hour), 2hour, 4hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  AUCt of Pioglitazone M-IV (Blood samples are collected 14 times for eachour Period.)
Pharmacokinetic variables - Cmax of Pioglitazone M-IV | Pre-dose (0hour), 2hour, 4hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  Cmax of Pioglitazone M-IV (Blood samples are collected 14 times for eachour Period.)
Pharmacokinetic variables - AUC∞ of Pioglitazone M-IV | Pre-dose (0hour), 2hour, 4hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  AUC∞ of Pioglitazone M-IV (Blood samples are collected 14 times for eachour Period.)
Pharmacokinetic variables - AUCt/AUC∞ of Pioglitazone M-IV | Pre-dose (0hour), 2hour, 4hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  AUCt/AUC∞ of Pioglitazone M-IV (Blood samples are collected 14 times for eachour Period.)
Pharmacokinetic variables - Tmax of Pioglitazone M-IV | Pre-dose (0hour), 2hour, 4hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  Tmax of Pioglitazone M-IV (Blood samples are collected 14 times for eachour Period.)
Pharmacokinetic variables - t1/2 of Pioglitazone M-IV | Pre-dose (0hour), 2hour, 4hour, 6hour, 8hour, 10hour, 12hour, 14hour, 16hour, 18hour, 24hour, 48hour, 72hour, 96hour
  t1/2 of Pioglitazone M-IV (Blood samples are collected 14 times for eachour Period.)

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, Gwanakgu, South Korea

IPD SHARING:
Plan to Share IPD: No